# **Statistical Analysis Plan**

A Randomized, Double-Blind, Placebo-Controlled, Parallel Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Estradiol Vaginal Cream USP, 0.01% (Teva Pharmaceuticals, USA) to Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott) in the Treatment of Atrophic Vaginitis

**Study Number 71436001** 

NCT03294538

Statistical Analysis Plan Approval Date: 04 August 2016

A Randomized, Double-Blind, Placebo-Controlled, Parallel Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Estradiol Vaginal Cream USP, 0.01% (Teva Pharmaceuticals, USA) to Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott) in the Treatment of Atrophic Vaginitis

Protocol Number: 71436001 Study Number: 71436001

#### **Sponsor:**

Teva Pharmaceuticals, USA 1090 Horsham Rd North Wales, PA 19454

**Contract Research Organization:** 

August 4, 2016

Final Version 1.0

# SAP FINAL VERSION APPROVALS

A Randomized, Double-Blind, Placebo-Controlled, Parallel Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Estradiol Vaginal Cream USP, 0.01% (Teva Pharmaceuticals, USA) to Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott) in the Treatment of Atrophic Vaginitis

| Written By: | |
|---------------------------|-------|
| Signature: | Date: |
| Reviewed By: | |
| Signature: | Date: |
| Approved By: | |
| Signature: | Date: |
| Teva Pharmaceuticals, USA | |

# Estradiol Vaginal Cream USP, 0.01%

# Protocol/Study Number 71436001

# **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|---|---|---|---|
| Draft 1.0 | July 25, 2016 | New Document | |
| Final 1.0 | August 4, 2016 | Incorporate client comments and finalize SAP | |

#### Estradiol Vaginal Cream USP, 0.01%

#### Protocol/Study Number 71436001

#### List of Abbreviations and Definition of Terms

ADaM Analysis Data Model

AE Adverse Event

C Celsius

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval CRF Case Report Form

CRO Contract Research Organization

dL Deciliter
F Fahrenheit

FDA Food & Drug Administration FSH Follicle-stimulating hormone

Hg Mercury

ICF Informed Consent Form

ICH International Conference on Harmonisation

LOCF Last Observation Carried Forward

mcg Microgram

MedDRA Medical Dictionary for Regulatory Activities

mg Milligram

mITT modified Intent-to-Treat Population

mL Milliliter mm Millimeter

OGD Office of Generic Drugs

PAP Papanicolaou

Measure of acidity/alkalinity рН PPP Per-Protocol Population Reference Listed Drug **RLD** SAE Serious Adverse Event SAP Statistical Analysis Plan SAS Statistical Analysis Software Study Data Tabulation Model **SDTM** United States of America U.S.A

# **TABLE OF CONTENTS**

| 1. | INTRODUCTION | 7 |
|---|---|---|
| 2. | OBJECTIVES | 7 |
| 3. | OVERALL STUDY DESIGN | 7 |
| 4. | RANDOMIZATION AND BLINDING | 10 |
| 5. | SAMPLE SIZE | 10 |
| 6. | ANALYSIS POPULATION | 11 |
| | STUDY ENDPOINTS | |
| 8. | STATISTICAL ANALYSIS METHODS | 12 |
| | 8.1 Baseline Characteristics | 12 |
| | 8.1.1 Patient Disposition | 12 |
| | 8.1.2 Demographic and Other Baseline Characteristics | |
| | 8.1.3 Medical History | 13 |
| | 8.1.4 Concomitant Medications | |
| | 8.1.5 Physical Exam | 14 |
| | 8.1.6 Laboratory Evaluations | 14 |
| | 8.1.7 Dosing Compliance | |
| | 8.2 Efficacy Analyses | 14 |
| | 8.2.1 Analysis of Primary Efficacy Endpoint | 15 |
| | 8.2.2 Analysis of Secondary Efficacy Endpoint | 16 |
| | 8.3 Safety Analysis | |
| | 8.3.1 Adverse Events | 17 |
| | 8.3.2 Vital Signs | 18 |
| | 8.4 Statistical Analysis Issues | 18 |
| | 8.5 Multiple Comparisons | 18 |
| | 8.6 Methods for Handling Missing Data | 18 |
| | 8.7 Interim Analyses | |
| 9. | TABLE, LISTING AND FIGURE SHELLS | 18 |
| | T16.1.9.1 Summary of Discontinued Patients | |
| | T16.1.9.2 Summary of Protocol Deviations (Safety Population) | 22 |
| | T16.1.9.3.1 Summary of Patients Excluded from Efficacy Analysis (Population | |
| | Determination) | 23 |
| | T16.1.9.3.2 Summary of Patients Included in Analysis Population by Study Center | 24 |
| | T16.1.9.4 Summary of Baseline Demographic Data (Safety Population) | 25 |
| | T16.1.9.5 Summary of Baseline Demographic Data (modified Intent-to-Treat | |
| | Population) | |
| | T16.1.9.6 Summary of Baseline Demographic Data (Per-Protocol Population) | 30 |
| | T16.1.9.7 Summary of Analysis Results of Primary Efficacy Endpoint (Proportion of | |
| | Responders Between Treatment Groups) | 31 |
| | T16.1.9.8 Summary of Analysis Results of Secondary Efficacy Endpoint (Proportion | |
| | of Treatment Successes Between Treatment Groups) | 32 |
| | T16.1.9.9 Overall Summary of Adverse Events (Safety Population) | 33 |

# Estradiol Vaginal Cream USP, 0.01% Protocol/Study Number 71436001

| T16.1.9.10.1 Summary of Frequency of All Adverse Events by Body System (Safet | ty |
|---|---|
| Population) | 34 |
| T16.1.9.10.2 Summary of Frequency for AEs Occurring in at Least 1% of Subjects | by |
| Body System (Safety Population) | 34 |
| T16.1.9.11 Summary of Frequency of All Adverse Events by Severity (Safety | |
| Population) | 35 |
| T16.1.9.12 Summary of Frequency of All Adverse Events by Relationship (Safety | |
| Population) | 36 |
| T16.1.9.13 Summary of Frequency of Serious Adverse Events (Safety Population). | 37 |
| T16.1.9.14 Summary of Adverse Events by Treatment (Safety Population) | 38 |
| T16.1.9.15 Summary of Vital Signs (Safety Population) | 39 |
| L16.2.1 Listing of Discontinued Patients | |
| L16.2.2 Listing of Protocol Deviations | 41 |
| L16.2.3.1 Patients Excluded from the Per-Protocol Population | 42 |
| L16.2.3.2 Patients Excluded from the Modified Intent-to-Treat Population | 43 |
| L16.2.4.1 Listing of Demographic Data | |
| L16.2.4.2 Listing of Patient Characteristics (Baseline Signs and Symptoms) | 45 |
| L16.2.4.3 Listing of Medical History | 46 |
| L16.2.4.4 Listing of Concomitant Medications | 47 |
| L16.2.5.1 Listing of Visit Date Information | 48 |
| L16.2.5.2 Listing of Drug Administration | 49 |
| L16.2.5.3 Listing of Study Compliance | |
| L16.2.6.1 Listing of Vaginal Cytology Results | 51 |
| L16.2.6.2 Listing of Signs and Symptoms Ratings | 52 |
| L16.2.7 Listing of Adverse Events by Treatment Group | 53 |
| L16.2.8.1 Listing of Laboratory Measurements | 54 |
| L16.2.8.2 Listing of Vaginal Ultrasonography and Mammogram | 55 |
| L16.2.8.3 Listing of Vital Signs | |
| 10. APPENDICIES | 58 |

#### Estradiol Vaginal Cream USP, 0.01%

Protocol/Study Number 71436001

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol 71436001 (Rev 0) dated 02-11-2015. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol 71436001 (Rev 0) dated 02-11-2015
- Case Report Form Booklet Version 1.0 for Study No. 71436001

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

#### 2. OBJECTIVES

- 1. Evaluate the therapeutic equivalence of the Test formulation, Estradiol Vaginal Cream USP, 0.01% (Teva Pharmaceuticals, USA) to the marketed product, Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott) in patients with atrophic vaginitis.
- 2. Demonstrate the superiority of the Test and Reference (active) treatments over Placebo (vehicle) cream in patients with atrophic vaginitis.
- 3. Compare the safety of Test, Reference and Placebo treatments in patients with atrophic vaginitis.

#### 3. OVERALL STUDY DESIGN

This randomized, double-blind, placebo-controlled, parallel group, multi-site study has been designed to evaluate the therapeutic efficacy and safety of a generic Estradiol Vaginal Cream USP, 0.01% (Teva Pharmaceuticals, USA) compared to the FDA Reference Listed Drug (RLD), Estrace<sup>®</sup> Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott) in patients with atrophic vaginitis. Additionally, both the Test and Reference products will be tested for superiority against a Placebo.

#### Estradiol Vaginal Cream USP, 0.01%

#### Protocol/Study Number 71436001

Following the 14-day screening period, patients who continue to meet the inclusion/exclusion criteria will be randomized in a 2:2:1 ratio (Test: Reference: Placebo) for 7 days of treatment. Up to 660 eligible postmenopausal female patients with atrophic vaginitis will be randomized, to obtain a mITT population with an estimated 250 patients in each of the active treatment groups and 125 in the Placebo treatment group.

Before any study-specific procedures are performed, all patients will read and sign the IRB-approved informed consent document.

To qualify for inclusion in the study, patients must be between the ages of 30-75 inclusive, postmenopausal with atrophic vaginitis assessed as moderate to severe using vaginal cytology, vaginal pH and patient-rated signs and symptoms. Patients cannot currently be undergoing treatment for atrophic vaginitis. Patients will only be eligible to participate in the study on one occasion and cannot have participated in another clinical research study within 30 days of being screened for this study.

At Visit 2 (Randomization), each qualified patient will be randomly assigned to one of the following treatment groups in a 2:2:1 ratio:

- Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)
- Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)
- Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Study medication will be self-administered by the patient for 7 days according to the dosing instructions provided. Each patient will be required to dose once a day at approximately the same time of day for 7 consecutive days.

During the study patients will visit the research center for a total of 3 scheduled visits:

- Visit 1/Screening (Day -14 to Day -1)
- Visit 2/Randomization (Day 1)
- Visit 3/End of Study (Day 8± 1)

Vaginal cytology and vaginal pH determination will be performed as a part of clinical evaluation at Visits 1 and 3. Visit 3 is to be scheduled on the day following the last day of dosing.

The primary efficacy endpoint is the proportion of patients in the per protocol (PP) population that are identified as "Responders" at the end of the treatment period evaluated on Day  $8 \pm 1$ . A responder is defined as a patient with at least a 25% reduction from baseline in the sum of % basal/parabasal + % intermediate cells on vaginal cytology AND vaginal pH < 5.0 with a change from baseline vaginal pH of at least 0.5.

# Estradiol Vaginal Cream USP, 0.01%

# Protocol/Study Number 71436001

# **Study Schematic**

| | Visit 1 | Visit 2 | Visit 3 |
|---|---|---|---|
| | Screening | Randomization | End of Study |
| | (Day -14 to Day-1) | (Day 1) | (Day $8 \pm 1$ ) or Early |
| | | | Termination |
| Informed Consent | X | | |
| Demographics | X | | |
| Medical History | X | X | |
| Inclusion/Exclusion<br>Criteria Review | X | X | |
| Vital Signs | X | X | X |
| Rating of Symptoms | X | X | X |
| Physical Exam Including<br>Pelvic Exam | X | | X |
| Breast Exam | X | | |
| Vaginal Cytology and pH | X | | X |
| PAP* | X | | |
| Serum FSH, Fasting<br>Triglycerides | X | | |
| Mammogram** | X | | |
| Vaginal Ultrasound*** | X | | |
| Dispense/Collect<br>Study Medication | | X | X |
| Dispense, Collect,<br>Review Patient Diary | | X | X |
| Adverse Events | | | X |
| Concomitant Medications | X | X | X |

<sup>\*</sup> Patients who do not have documentation of a PAP smear completed within the last 12 months.

<sup>\*\*</sup>Patients over the age of 40 who do not have documentation of a mammogram completed within the 9 months before screening will have a mammogram as part of the screening evaluations.

<sup>\*\*\*</sup>Patients with an intact uterus will have a vaginal ultrasound as part of the screening evaluations

# Estradiol Vaginal Cream USP, 0.01%

Protocol/Study Number 71436001

| 4. RANDOMIZATION AND BLINDING |
|---|
| The study drug will be randomized, packaged and blinded by an independent packaging company. Randomization will be pre-planned according to a computer-generated randomization |
| Each patient will be provided. |
| with one patient kit, containing 1 tube of study medication. |
| Each patient will receive a screening number at Visit 1, which will be recorded in the patient's CRF. At Visit 2, eligible patients will receive a randomization number (based on treatment assigned), which will be recorded in the CRF. |
| Patients will be randomized to a treatment regimen by assigning treatments in sequential order. At the end of the study, after all the clinical data has been entered and the study database has been locked, a copy of the randomization will be sent to the statistician. |
| The Investigator, staff at the study site, study monitors, and data analysis/management personnel will be blinded to the patient assignment. |
| 5. SAMPLE SIZE |
| The primary statistical analysis of interest is the proportion of patients in the Per Protocol (PP) population that are identified as "Responders" at the end of the treatment period evaluated on Day $8 \pm 1$ . |
| a sample size of 224 patients per active group in the PP population to demonstrate bioequivalence (i.e., the 90% confidence interval (Yates' continuity-corrected) of the absolute difference between the Test and Reference "Responder" rate rates is within a defined equivalence range [-20%, +20%]). |
| Using a 2:1 (active: placebo) randomization scheme, and assuming the conversion rate from mITT to PP will be about 90%, 250 patients in each of active groups and |
| 125 patients in the placebo group of the mITT population demonstrate superiority of active over placebo. |

To allow for about 5% of patients who may drop out from the study or are

#### Estradiol Vaginal Cream USP, 0.01%

#### Protocol/Study Number 71436001

otherwise non-evaluable, up to 660 patients may be randomized to obtain 625 patients in the mITT population (i.e., 250 in each active group and 125 in the Placebo group).

#### 6. ANALYSIS POPULATION

# Per-Protocol (PP) Population

Patients will be eligible for inclusion in the PP population if they:

- Met the inclusion/exclusion criteria as defined in the protocol at Visit 1 and 2
- Did not take any prohibited medications throughout the study
- Did not have any significant deviations from the protocol
- Did not develop any concurrent vaginal infection or illness exhibiting symptoms similar to atrophic vaginitis, or symptoms that in the Investigator's opinion would interfere with primary and secondary endpoint assessments
- Completed the last study visit (Visit 3) Day  $8 \pm 1$ .
- Were compliant with dosing between 75%-125% of the required doses (6 8 doses), and did not miss more than 1 dose
- Any patient who withdrew from the study because of lack of efficacy will be included
  in the PP population as a Non-Responder. Patients who discontinue early for other
  reasons should be excluded from the PP population and included in the mITT
  population using Last Observation Carried Forward (LOCF).

#### **Modified Intent-to-Treat (mITT) Population**

The mITT population will include all patients in the PP population, AND patients who:

- Administered at least one dose of randomized study medication and
- Had a post-randomization evaluation

#### **Safety Population**

The safety population will include all patients who are randomized and administered at least one dose of study drug.

#### 7. STUDY ENDPOINTS

#### Primary Efficacy Endpoint

#### Estradiol Vaginal Cream USP, 0.01%

#### Protocol/Study Number 71436001

The primary efficacy endpoint is the proportion of patients in the PP population that are identified as "Responders" at the end of the treatment period evaluated on Day  $8 \pm 1$ .

A responder is defined as a patient with at least a 25% reduction from baseline in the sum of % basal/parabasal + % intermediate cells on vaginal cytology AND vaginal pH < 5.0 with a change from baseline vaginal pH of at least 0.5.

#### Secondary Efficacy Endpoint

The secondary efficacy endpoint is the proportion of patients in the PP population that are identified as "Treatment Success" at the end of the treatment period evaluated on Day  $8 \pm 1$ .

A "Treatment Success" is defined as a score of 0 or 1 at Day  $8 \pm 1$  for the symptom identified at baseline as the most bothersome. This evaluation is to be based on patient self-assessed symptoms of vulvar and vaginal atrophy on a scale of 0 to 3 where 0 = none and 3 = severe.

#### 8. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p<0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics, efficacy variables and safety variables.

For categorical variables, the number and percent of each category within a parameter will be calculated for non-missing data. For continuous variables, statistics will include n, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS®, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model).

#### 8.1 Baseline Characteristics

#### 8.1.1 Patient Disposition

The patient accountability and disposition information will be summarized by study treatment group. The number of patients enrolled, randomized, and the number of patients in each analysis population will be tabulated. In addition, completion status and primary reason for withdrawal will be summarized by study treatment group.

#### Estradiol Vaginal Cream USP, 0.01%

## Protocol/Study Number 71436001

#### 8.1.2 Demographic and Other Baseline Characteristics

Baseline comparability of all treatment groups will be evaluated separately in the PP, mITT and Safety populations. The following baseline demographics (determined from their initial study visit) will be evaluated:

- Age (years)
- Gender (male/female)
- Ethnicity (Hispanic/non Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native, Other)
- natural or surgical menopause
- duration of postmenopausal status
- baseline signs and symptoms
- baseline % of the three major vaginal wall cell types (basal/parabasal cells, intermediate cells and superficial cells)
- vaginal pH

Summary tables by treatment group will be presented. Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, maximum).

Categorical variables will be summarized using frequencies and percentage. Baseline treatment comparisons will be presented using Cochran-Mantel-Haenszel test for the categorical variables, and Analysis of Variance for the continuous variables.

All data will be listed by treatment and patient.

#### **8.1.3 Medical History**

At Visit 1 patients will be questioned about medical history, including acute and chronic medical history and medical history relevant to their vaginal atrophy. At Visit 2 medical history will be reviewed and updated if changes have occurred.

Medical history data will be listed by treatment and patient.

#### **8.1.4 Concomitant Medications**

At Visit 1 patients will be questioned about all concomitant medication use within the previous 6 months.

#### Estradiol Vaginal Cream USP, 0.01%

#### **Protocol/Study Number 71436001**

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment and patient.

#### 8.1.5 Physical Exam

At Visit 1 the Investigator will perform a general physical exam including pelvic exam and breast exam. At Visit 3 the Investigator will perform a general physical exam including pelvic exam, any negative findings on exam should be reported as Adverse Events.

Physical examination results will be listed by treatment and patient.

#### 8.1.6 Laboratory Evaluations

All patients will have a blood sample taken for evaluation of serum FSH levels. Serum FSH will be evaluated by a central clinical laboratory. Patients must have a Serum FSH > 40mIU/ml to be eligible for participation in the study.

All patients will have a blood sample taken for fasting triglyceride testing. These samples will be sent to the central laboratory for testing. Patients with fasting triglyceride values > 350 mg/dL will not be eligible for inclusion in the study.

Laboratory evaluation results will be listed by treatment and patient.

# **8.1.7 Dosing Compliance**

Dosing compliance will be checked by site staff at Visit 3 by reviewing patient diary entries. Patients will be considered compliant with dosing if they administer 75% - 125% of the required number of doses, and do not miss more than 1 dose.

Drug administration and dosing compliance will be listed by treatment and patient.

#### 8.2 Efficacy Analyses

The following symptoms (see Appendix A for detailed rating scales) will be evaluated at Visits 1, 2 and 3 by the blinded clinical staff or Investigator.

| Symptoms | Rating Scales |
|---|---|
| Vaginal Dryness | 0=None, 1=mild, 2=moderate, 3=severe |
| Vaginal/Vulvar irritation/itching | 0=None, 1=mild, 2=moderate, 3=severe |
| Dysuria | 0=None, 1=mild, 2=moderate, 3=severe |
| Vaginal Pain associated with Sexual Activity | 0=None, 1=mild, 2=moderate, 3=severe |
| Vaginal Bleeding | 0= Absent, 1= Present |

The patients will be asked to identify which symptom is considered to be the most bothersome symptom at Visit 1 and Visit 2. Vaginal Pain associated with Sexual Activity or Vaginal

#### Estradiol Vaginal Cream USP, 0.01%

#### Protocol/Study Number 71436001

Bleeding are acceptable to be considered most bothersome symptom only if patient is currently sexually active and plans to remain so throughout the study.

#### 8.2.1 Analysis of Primary Efficacy Endpoint

#### Therapeutic Bioequivalence Analysis

Therapeutic equivalence of the Test product to the Reference product based on the primary endpoint will be evaluated in the PP population after the end of treatment on Day  $8 \pm 1$ .

Based on the usual method used in OGD for binary outcomes, the 90% confidence interval for the difference in success proportions between test and reference treatment should be contained within [-0.20, +0.20] in order to establish equivalence.

The compound hypothesis to be tested is:

$$H_0: P_T - P_R < -.20 \text{ or } P_T - P_R > .20 \text{ versus}$$

$$H_A: -.20 \le P_T - P_R \le .20$$

where  $P_T$  = cure rate of test treatment

 $P_R$  = cure rate of reference treatment.

Let

 $n_T$  = sample size of test treatment group

 $cn_T$  = number of cured patients in test treatment group

 $n_R$  = sample size of reference treatment group

 $cn_R$ = number of cured patients in reference treatment group

$$\hat{P}_T = c n_T / n_T$$
  $\hat{P}_R = c n_R / n_R$ , and

$$se = (\hat{P}_T (1 - \hat{P}_T)/n_T + \hat{P}_R (1 - \hat{P}_R)/n_R)^{1/2}$$

The 90% confidence interval for the difference in proportions between test and reference will be calculated as follows, using Yates' correction:

$$L = (\hat{P}_T - \hat{P}_R) - 1.645 se - (1/n_T + 1/n_R)/2$$

$$U = (\hat{P}_T - \hat{P}_R) + 1.645 se + (1/n_T + 1/n_R)/2$$

If the 90% confidence interval (calculated using Yates' continuity correction) for the absolute

#### Estradiol Vaginal Cream USP, 0.01%

Protocol/Study Number 71436001

difference between the proportion of patients considered as "Responders" (at least a 25% reduction from baseline in the sum of % basal/parabasal + % intermediate cells on vaginal cytology AND vaginal pH < 5.0 with a change from baseline vaginal pH of at least 0.5) in the Test and Reference groups is contained within the range [-20%, +20%] then bioequivalence of the Test product to the Reference product will be considered to have been demonstrated for the primary endpoint.

## **Superiority to Placebo Analysis**

The mITT population and LOCF will be used to evaluate the superiority of both the Test and Reference product to Placebo.

For the determination of superiority the proportion of patients who are considered as "Responders" in the test and reference product groups will each be compared to the proportion of "Responders" in the placebo product group. On condition that both the test and the reference group demonstrate statistically greater proportion of "Responders" (p< 0.05, 2-sided) than the placebo group then superiority shall be concluded and the sensitivity of the methodology confirmed.

Summary table with frequency and percentage on the proportion of responders by treatment group will be presented. Treatment comparison for Test vs. Placebo and Reference vs. Placebo will be performed by continuity-corrected Z-tests. The superiority of Test and Reference treatments over the Placebo will be evaluated identically in separate Z-Test analyses.

#### 8.2.2 Analysis of Secondary Efficacy Endpoint

#### **Therapeutic Bioequivalence Analysis**

Similar to the analysis for primary endpoint above, therapeutic equivalence of the Test product to the Reference product based on the secondary endpoint will be evaluated in the PP population after the end of treatment on Day  $8 \pm 1$ .

Secondary analysis will compare the proportion of patients considered to be a "Treatment Success" for their most bothersome symptom. A "Treatment Success" is defined as a score of 0 or 1 at Day 8 for the symptom identified at baseline as the most bothersome). If the 90% confidence interval (calculated using Yates' continuity correction) for the absolute difference between the proportion of patients considered as "Treatment Success" in the Test and Reference groups is contained within the range [-20%, +20%] then bioequivalence of the Test product to the Reference product will be considered to have been demonstrated for the secondary endpoint.

To declare therapeutic equivalence of the Test product to the Reference product, bioequivalence

#### Estradiol Vaginal Cream USP, 0.01%

#### Protocol/Study Number 71436001

must be demonstrated for only the primary endpoint. Bioequivalence testing of the secondary endpoint will be conducted for supportive information.

#### **Superiority to Placebo Analysis**

The mITT population and LOCF will be used to evaluate the superiority of both the Test and Reference product to Placebo.

Similar to the analysis for primary endpoint above, superiority of the Test and Reference products against the Placebo for secondary endpoints will be tested at the 5% significance level (p < 0.05; using two-sided, continuity-corrected Z-test) in the mITT population using last observation carried forward. The superiority of Test and Reference treatments over the Placebo will be evaluated identically in separate Z-Test analyses.

#### 8.3 Safety Analysis

#### 8.3.1 Adverse Events

All the adverse events (AEs) reported will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 17.0 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

All AEs will be listed by patient and treatment.

The total number and percentage of patients with at least one AEs, discontinued study drug due to AEs, AE severity and AEs related to investigational product, serious AEs and death will be summarized by treatment groups and overall.

A summary table of the number and percent of patients with AEs by system organ class, preferred term, and treatment group will be presented. Each patient will be counted only once within each preferred term.

A frequency summary table of the number of AEs by system organ class, preferred term, severity, and treatment group will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug, and treatment group will be presented. Relationship to a study drug will be classified as "Related" or "Not Related".

Should sufficient data exist, adverse event frequencies will be compared between treatments using the Chi-square testing (Fisher's exact test if appropriate).

#### Estradiol Vaginal Cream USP, 0.01%

Protocol/Study Number 71436001

#### 8.3.2 Vital Signs

The patient's vital signs will be recorded (pulse, blood pressure, temperature and respiration rate) at Visits 1, 2, and 3 or end of study.

Descriptive summaries (n, mean, standard deviation, minimum, median and maximum) will be provided by treatment and visit. The summary table will be based on safety population randomized.

All data will be listed by treatment and patient.

#### **8.4 Statistical Analysis Issues**

As this is a multiple-site study, treatment-by-site interaction analysis will be examined using the Cochran-Mantel-Haenszel Test for the primary efficacy variable, the proportion of patients in the PPP that are considered to be a "responder" at Visit 3. A site(s) with a low enrollment rate(s) may be pooled with its geographically closest site. The pooling will be done for low enrolling sites that account for less than 4-7% of the total number of patients in the PP population (equivalence test) and mITT population (superiority tests) at the site with the highest enrolling rate.

#### 8.5 Multiple Comparisons

No multiple comparison adjustment will be made in this study.

#### 8.6 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Patients with missing data will be excluded only from analyses for which data are not available.

Any patient who withdrew from the study because of lack of efficacy will be included in the PP population as a Non-Responder. Patients who discontinue early for other reasons should be excluded from the PP population and included in the mITT population using Last Observation Carried Forward (LOCF).

#### 8.7 Interim Analyses

There is no interim analysis planned in this study.

#### 9. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to

# Estradiol Vaginal Cream USP, 0.01%

# Protocol/Study Number 71436001

show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

TABLE, LISTING AND FIGURE SHELLS

**T16.1.9.1 Summary of Discontinued Patients** 

| Patients | Test | Reference | Placebo | Total |
|--------------------------|------|-----------|---------|-------|
| Screened | | | | xxx |
| Screen failures | | | | xxx |
| Randomized | XXX | xxx | XXX | xxx |
| Completed Study | XXX | xxx | XXX | XXX |
| Terminated Early | xxx | xxx | xxx | xxx |
| Early Termination Reason | | | | |
| Adverse Event | xxx | XXX | XXX | xxx |
| Lack of efficacy | XXX | xxx | XXX | xxx |
| Lost to Follow-Up | xxx | xxx | xxx | xxx |
| etc. | | | | |

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies Sas Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.2 Summary of Protocol Deviations (Safety Population)

| | Test | Reference | Placebo | Total |
|---|---|---|---|---|
| Total Patients with Protocol Deviations | XXX | xxx | XXX | XXX |
| Total Deviations | xxx | xxx | xxx | XXX |
| Dosing Non-Compliance (Missed > one doses) | xxx | XXX | xxx | XXX |
| Failure to meet randomization criteria | XXX | xxx | XXX | XXX |
| Lost to Follow-up | xxx | xxx | xxx | XXX |
| Outside Visit Window | XXX | xxx | XXX | XXX |
| Patient Dosed on the Day of Visit 3 | XXX | XXX | XXX | XXX |
| Restricted Medication | XXX | xxx | XXX | XXX |
| Total Dosing Non-Compliance | XXX | XXX | XXX | XXX |
| Other | XXX | XXX | XXX | xxx |

Reference: Estrace<sup>®</sup> Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.3.1 Summary of Patients Excluded from Efficacy Analysis (Population Determination)

| | | Test | Reference | Placebo | Total |
|---|---|---|---|---|---|
| Randomized | Total | XXX | XXX | xxx | XXX |
| Safety Population | Total | XXX | XXX | XXX | XXX |
| Excluded from Safety | Did Not Dose | XXX | XXX | XXX | XXX |
| mITT Population | Total | XXX | xxx | xxx | XXX |
| Excluded from mITT | Inclusion/Exclusion | xxx | XXX | XXX | XXX |
| | etc. | | | | |
| PP Population | Total | XXX | xxx | XXX | XXX |
| Excluded from Excluded from PPP | Restricted Medication | xxx | XXX | XXX | XXX |
| | Outside of Visit 3 Window | | | | |
| | etc. | | | | |

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies Sas Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.3.2 Summary of Patients Included in Analysis Population by Study Center

| | | | | | PPP | | | | mITT | | | | Safety | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site<br>No. | Name | Total<br>Randomized | Test | Ref | Placebo | Total | Test | Ref | Placebo | Total | Test | Ref | Placebo | Total |
| XX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.4 Summary of Baseline Demographic Data (Safety Population)

| | | Test (N = xxx) | Reference $(N = xxx)$ | $ \begin{array}{l} Placebo \\ (N = xxx) \end{array} $ | P-value |
|---|---|---|---|---|---|
| Age (years) | n | XXX | xxx | xxx | x.xxxx |
| | Mean $\pm$ SD | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Race | American Indian or Alaska Native | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | X.XXXX |
| | Asian | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Black/African American | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Native Hawaiian or other Pacific Islander | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | White | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Gender | Female | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Male | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Ethnicity | Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Not Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm


T16.1.9.4 Summary of Baseline Demographic Data (Safety Population)

| | | Test (N = xxx) | Reference $(N = xxx)$ | $\begin{aligned} & \text{Placebo} \\ & (\text{N} = xxx) \end{aligned}$ | P-value |
|---|---|---|---|---|---|
| Natural or Surgical Menopause | Natural | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Surgical | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Vaginal Dryness | None | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Vaginal/Vulvar Irritation/Itching | None | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.4 Summary of Baseline Demographic Data (Safety Population)

| | | Test | Reference | Placebo | P-value |
|---|---|---|---|---|---|
| | | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | |
| Dysuria | None | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | X.XXXX |
| | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Vaginal Pain during Sexual Activity | None | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Most Bothersome Sign or Symptom | Vaginal Dryness | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Vaginal/Vulvar Irritation/Itching | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Dysuria | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Vaginal Pain during<br>Sexual Activity | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Vaginal Bleeding | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Created on: ddmmmyy hh:mm


T16.1.9.4 Summary of Baseline Demographic Data (Safety Population)

| | | Test | Reference | Placebo | P-value |
|---|---|---|---|---|---|
| | | (N = xxx) | (N = xxx) | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | |
| Vaginal Bleeding | Absent | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Present | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Duration of Postmenopausal<br>Status (Years) | XXX | XXX | xxx | xxx | |
| | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | x.xxxx |
| | XX.X | XX.X | XX.X | XX.X | |
| | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| % of basal/parabasal cells | XXX | XXX | XXX | XXX | |
| | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | X.XXXX |
| | XX.X | XX.X | XX.X | XX.X | |
| | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

 $Path: L: \Studies\_Sas\_Codes \Clinical\ Trial \71436001 \PDF \xxx$ 

Created on: ddmmmyy hh:mm


T16.1.9.4 Summary of Baseline Demographic Data (Safety Population)

| | | Test (N = xxx) | Reference $(N = xxx)$ | $ Placebo \\ (N = xxx) $ | P-value |
|---|---|---|---|---|---|
| % of intermediate cells | n | XXX | XXX | XXX | X.XXXX |
| | $Mean \pm SD$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | |
| | Median | XX.X | xx.x | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| % of superficial cells | n | XXX | XXX | XXX | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | |
| | Median | xx.x | xx.x | xx.x | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Vaginal pH | n | XXX | XXX | XXX | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | $xx.x \pm xx.xx$ | |
| | Median | xx.x | XX.X | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Created on: ddmmmyy hh:mm

08/04/2016

Similar tables will be created for T16.1.9.5 and T16.1.9.6

T16.1.9.5 Summary of Baseline Demographic Data (modified Intent-to-Treat Population)

T16.1.9.6 Summary of Baseline Demographic Data (Per-Protocol Population)

T16.1.9.7 Summary of Analysis Results of Primary Efficacy Endpoint (Proportion of Responders Between Treatment Groups)

**Equivalence: Per-Protocol Population** 

| | | | | <b>Difference Between Treatments</b> | |
|---|---|---|---|---|---|
| Treatment | Number of | Number of | <b>Proportion of</b> | | |
| Group | Patients (N) | Responders (n) | Responders (%) | Difference | 90% CI Evaluation |
| Test | XXX | XXX | XX.X <sup>0</sup> / <sub>0</sub> | | |
| Reference | XXX | XXX | XX.X <sup>0</sup> / <sub>0</sub> | XX.X% | xx.x - xx.x |

**Superiority: modified Intent-to-Treat Population** 

| | | | | Treatment | vs. Placebo |
|---|---|---|---|---|---|
| Treatment | Number of | Number of | Proportion of | | |
| Group | Patients (N) | Responders (n) | Responders (%) | Difference | P-value |
| Placebo | xxx | xxx | xx.x% | | |
| Test | xxx | xxx | xx.x% | xx.x% | x.xxxx |
| Placebo | xxx | xxx | xx.x% | | |
| Reference | xxx | xxx | xx.x% | xx.x% | x.xxxx |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

# T16.1.9.8 Summary of Analysis Results of Secondary Efficacy Endpoint (Proportion of Treatment Successes Between Treatment Groups)

**Equivalence: Per-Protocol Population** 

| - | | | | <b>Difference Between Treatments</b> | |
|---|---|---|---|---|---|
| Treatment<br>Group | Number of<br>Patients (N) | Number of<br>Treatment<br>Successes (n) | Proportion of<br>Treatment<br>Successes (%) | Difference | 90% CI Evaluation |
| Test | xxx | XXX | XX.X <sup>0</sup> / <sub>0</sub> | | |
| Reference | xxx | xxx | xx.x% | xx.x% | xx.x - xx.x |

**Superiority: modified Intent-to-Treat Population** 

| Treatment<br>Group | | Number of | Proportion of | Treatment | vs. Placebo |
|---|---|---|---|---|---|
| | Number of Patients (N) | Treatment Successes (n) | Treatment Successes (%) | Difference | P-value |
| Placebo | xxx | XXX | XX.X% | | |
| Test | XXX | XXX | xx.x% | xx.x% | X.XXXX |
| Placebo | XXX | XXX | xx.x% | | |
| Reference | XXX | XXX | XX.X% | xx.x% | x.xxxx |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.9 Overall Summary of Adverse Events (Safety Population)

| Description | Test<br>N (%) | Reference<br>N (%) | Placebo<br>N (%) | Total<br>N (%) |
|---|---|---|---|---|
| Patients Randomized | XXX | XXX | XXX | XXX |
| Patients with at least one AE | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Discontinued study drug due to above AE | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| AEs reported | xxx | XXX | XXX | xxx |
| Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Not Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Related | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Death | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Serious AE | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

Related = Probable, Possible, Unlikely

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies Sas Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

T16.1.9.10.1 Summary of Frequency of All Adverse Events by Body System (Safety Population)

| | Test $(N = xxx)$ | | Reference (N = xxx) | | $ Placebo \\ (N = xxx) $ | | Fisher's | |
|---|---|---|---|---|---|---|---|---|
| <b>Body System</b> | MedDRA Term | Events | Patients | Events | Patients | Events | Patients | P-value |
| Patients with at least one AE | Total | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | x.xxxx |
| Ear and labyrinth disorders | Ear pain | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | x.xxxx |
| | etc. | | | | | | | |

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Comparison of treatment groups is with respect to the number of patients with at least one occurrence of the AE.

Path: L:\Studies Sas Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm


Similar Table will be created for:

T16.1.9.10.2 Summary of Frequency for AEs Occurring in at Least 1% of Subjects by Body System (Safety Population)

T16.1.9.11 Summary of Frequency of All Adverse Events by Severity (Safety Population)

| | | | Test # of Events (N=xx) | | | Reference<br># of Events<br>(N=xx) | | | Placebo<br># of Events<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Body System | MedDRA Term | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Total AEs | Total | xx(xx.x%) | xx(xxx%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xxx%) | xx(xxx%) |
| Ear and labyrinth disorders | Earpain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xxx%) | xx (xx.x%) | xx (xx.x%) | xx(xxx%) | xx (xx.x%) | xx (xx.x%) |
| | Hypoacusis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

N = Total number of events in each treatment group; Percentage is based on total number of events.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm
T16.1.9.12 Summary of Frequency of All Adverse Events by Relationship (Safety Population)

| | | Test # of Events (N=xx) | | #of I | erence<br>Events<br>=xx) | #of1 | cebo<br>Events<br>=xx) |
|---|---|---|---|---|---|---|---|
| Body System | MedDRA Term | Related | Not Related | Related | Not Related | Related | Not Related |
| Total AEs | Total | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xxx%) |
| Ear and labyrinth disorders | Earpain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) |
| | Hypoacusis | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

N = Total number of events in each treatment group; Percentage is based on total number of events.

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

# T16.1.9.13 Summary of Frequency of Serious Adverse Events (Safety Population)

| Body System | MedDRA Term | Test<br># Events | Reference<br># Events | Placebo<br># Events |
|---|---|---|---|---|
| Injury, poisoning and procedural complications | Alcohol poisoning | XX | XX | XX |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

# T16.1.9.14 Summary of Adverse Events by Treatment (Safety Population)

Test: Estradiol Vaginal Cream, USP, 0.01%

| | | Severity | | | |
|---|---|---|---|---|---|
| Body System<br>MedDRA Term | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Related<br>n (%) | Not Related<br>n (%) |
| Total AEs (N=xxx) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Ear and labyrinth disorders Hypoacusis etc. | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) | xx ( xx.x%)<br>xx ( xx.x%) |
| etc. | | | | | |

N = Total AEs in Test Group

n (%) = Number of AEs (Percent of Total AEs in Test Group)

Path: L:\Studies Sas Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

Note to programmer: Similar tables will be created for Reference and Placebo groups.

T16.1.9.15 Summary of Vital Signs (Safety Population)

| Vital Signs | Visit | Statistic | Test (N = xxx) | Reference $(N = xxx)$ | $\begin{aligned} & \textbf{Placebo} \\ & (\textbf{N} = \textbf{x} \textbf{x}) \end{aligned}$ |
|---|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | 1 | n | XXX | XXX | xxx |
| | | $Mean \pm SD$ | $xxx.x \pm xx.xx$ | $xxx.x \pm xx.xx$ | $xxx.x \pm xx.xx$ |
| | | Median | XXX.X | xxx.x | xxx.x |
| | | Range | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| | 2 | | | | |
| | 3 | | | | |

Diastolic Blood Pressure (mmHg)

Heart Rate (beats/min)

Respiration Rate (breaths/min)

Temperature (F)

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

#### L16.2.1 Listing of Discontinued Patients

| Treatment<br>Group | Patient<br>Randomization<br>Number | Discontinuation<br>Reason | Population |
|---|---|---|---|
| Test | XX-XXXX | Withdrew Consent | Per-Protocol |
| | XX-XXXX | Lost to Follow-up | Safety |

Reference Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies Sas Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

#### L16.2.2 Listing of Protocol Deviations

| Treatment<br>Group | Patient<br>Randomization<br>Number | <b>Event Description</b> | Population |
|---|---|---|---|
| Test | XX-XXXX | Outside Visit Window (Visit: 3) | Per-Protocol |

Reference Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

# L16.2.3.1 Patients Excluded from the Per-Protocol Population

| Treatment<br>Group | Patient<br>Randomization<br>Number | Exclusion Reason |
|---|---|---|
| Test | XX-XXXX | Patient did not meet IE criterion |
| | XX-XXXX | Patient took prohibited medications |
| Reference<br>Placebo | | |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

#### L16.2.3.2 Patients Excluded from the Modified Intent-to-Treat Population

| Treatment<br>Group | Patient<br>Randomization<br>Number | Exclusion Reason |
|---|---|---|
| Test | XX-XXXX | Patient did not have at least one post-randomization evaluation |

Reference Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm


# L16.2.4.1 Listing of Demographic Data

| Treatment<br>Group | Patient<br>Randomization<br>Number | Age<br>(years) | Gender | Ethnicity | Race | Natural or Surgical<br>Menopause |
|---|---|---|---|---|---|---|
| Test | xx-xxxx | 30 | Female | Not Hispanic or Latino | Black or African American | Natural |
| | | | | Surgical | | |

Reference

Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies Sas Codes\Clinical Trial\71436001\PDF\xxx

#### L16.2.4.2 Listing of Patient Characteristics (Baseline Signs and Symptoms)

| | | | Ba | seline Signs | and Symptoms S | Scores | | | Baseline | % | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Patient<br>Rando-<br>mization<br>Number | Vaginal<br>Dryness | Vaginal/<br>Vulvar<br>Irritation/<br>itching | Dysuria | Vaginal Pain<br>Associated<br>With Sexual<br>Activity | Vaginal<br>Bleeding | Most<br>Bothersome<br>Symptom<br>(Baseline) | Superficial<br>Cells | Basal/<br>para<br>Basal<br>Cells | Intermediate<br>Cells | Baseline<br>Vaginal<br>pH |
| Test | XX-XXXX | 1 | 2 | 2 | 2 | 1 | Vaginal<br>Dryness | 6 | 0 | 94 | 5.5 |

Reference

Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace<sup>®</sup> Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

#### L16.2.4.3 Listing of Medical History

| Treatment<br>Group | Patient<br>Randomization<br>Number | System | Diagnosis or Surgical<br>Procedure | Start Date | End Date | Ongoing |
|---|---|---|---|---|---|---|
| Test | XX-XXXX | Gynecologic | Menopause | 2003 | 2003 | |

Reference Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

### L16.2.4.4 Listing of Concomitant Medications

| Treatment<br>Group | Patient<br>Randomization<br>Number | Treatment<br>Area | Medication | Dosage | Frequency | Route | Start/End<br>Date | Indication |
|---|---|---|---|---|---|---|---|---|
| Test | xx-xxxx | Yes | LISINOPRIL | 20 MG | QD | РО | yyyy-mm-dd/<br>yyyy-mm-dd | HYPERTENSION |

Reference Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

#### L16.2.5.1 Listing of Visit Date Information

| | Patient | | | | _ |
|---|---|---|---|---|---|
| Treatment | Randomization | <b>Informed Consent</b> | | | Visit 3 or |
| Group | Number | Date | Visit 1 | Visit 2 | <b>Early Termination</b> |
| Test | xx-xxxx | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd |

Reference

Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

#### L16.2.5.2 Listing of Drug Administration

| Treatment<br>Group | Patient<br>Randomization<br>Number | Date of<br>First Dose | Date of<br>Last Dose | Total Number of Dose Administered | Dosing<br>Compliance<br>(%) |
|---|---|---|---|---|---|
| Test | XX-XXXX | yyyy-mm-dd | yyyy-mm-dd | XX | XXX.X |

Reference Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

# L16.2.5.3 Listing of Study Compliance

| Treatment<br>Group | Patient<br>Randomi-<br>zation<br>Number | Dose on<br>the day of<br>Visit 3? | Use any restricted medication for the treatment of atrophic vaginitis? | Use any restricted medication other than for the treatment of atrophic vaginitis? | Administer < 6 or >8 of the intended doses? | Miss >1<br>dose<br>of study<br>medication? | Develop any concurrent vaginal infection or illness? | Require additional treatment? |
|---|---|---|---|---|---|---|---|---|
| Test | XX-XXXX | No | No | No | No | No | No | No |

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

# L16.2.6.1 Listing of Vaginal Cytology Results (Test: Estradiol Vaginal Cream, USP, 0.01%)

| | Baseline | | | Visit 3 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>Rando-<br>mization | Basal/<br>Parabasal | Inter-<br>mediate | Basal/<br>Parabasal<br>+Inter- | Super-<br>ficial | | Basal/<br>Parabasal | Inter-<br>mediate | Basal/<br>Parabasal<br>+Inter- | Super-<br>ficial | | Cytology<br>Changes<br>From | pH<br>Changes<br>From | Responder |
| Number | % | % | mediate% | Cells% | pН | % | % | mediate% | Cells% | pН | Baseline | Baseline | Yes/No |
| xx-xxxx | 69 | 31 | 100 | 100 | 7.0 | 12 | 43 | 55 | 100 | 4.5 | 45 | 2.5 | Yes |

Programming note: table will continue for reference and placebo group

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx


# L16.2.6.2 Listing of Signs and Symptoms Ratings

| | Patient | | | <b>Baseline Most</b> | |
|---|---|---|---|---|---|
| Treatment | Randomization | <b>Most Bothersome</b> | <b>Most Bothersome</b> | Bothersome | Success |
| Group | Number | Symptom at Baseline | Score at Baseline | Symptom Score at V3 | (Yes/No) |
| Test | XX-XXXX | Vaginal Dryness | 3 | 0 | Yes |

Reference

Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies Sas Codes\Clinical Trial\71436001\PDF\xxx

#### L16.2.7 Listing of Adverse Events by Treatment Group

| Treatment<br>group | Patient<br>Rando-<br>mization<br>Number | Body System/<br>MedDRA Term/<br>AE Term | Treatment<br>Area | End Date | Severity | Relationship to<br>Study Drug | Outcome | Action<br>Taken | Other<br>Action<br>Taken | SAE? |
|---|---|---|---|---|---|---|---|---|---|---|
| Test | xx-xxxx | NERVOUS SYSTEM<br>DISORDERS/ HEADACHE/<br>HEADACHE | Yes | yyyy-mm-dd/<br>yyyy-mm-dd | Mild | Not Related | Recovered | None | None | No |

Reference

Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

08/04/2016

### L16.2.8.1 Listing of Laboratory Measurements

| | Patient | | | |
|---|---|---|---|---|
| Treatment<br>Group | Randomization<br>Number | Collection<br>Date | Baseline FSH (mIU/ml) | Baseline Triglycerides (mg/dL) |
| Test | XX-XXXX | yyyy-mm-dd | 99.0 | 76 |

Reference

Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

#### L16.2.8.2 Listing of Vaginal Ultrasonography and Mammogram

| | | Vagir | Mammogram | | |
|---|---|---|---|---|---|
| Treatment<br>Group | Patient<br>Randomization<br>Number | Does Patient Have a Collection Confirmed Inactive Uterine Date Lining of < 4 mm?* | | Collection Date | Are Screening Mammogram Results Normal?** |
| Test | XX-XXXX | yyyy-mm-dd | Yes | yyyy-mm-dd | Yes |
| | XX-XXXX | | N/A | | N/A |

Reference

Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Note: \* N/A = Patient has had a hysterectomy; \*\* N/A = patient is  $\leq 40$  years of age

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

L16.2.8.3 Listing of Vital Signs

| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit | Systolic BP (mmHg) | Diastolic BP (mmHg) | Heart Rate (beats/min ) | Respiration Rate (breaths/min) | Temperature<br>(F) |
|---|---|---|---|---|---|---|---|
| Test | XX-XXXX | 1 | 120 | 70 | 84 | 18 | 98.6 |
| | | 2 | 140 | 80 | 74 | 18 | 97 |
| | | 3/EOS | 130 | 87 | 74 | 18 | 99.2 |

Reference Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies Sas Codes\Clinical Trial\71436001\PDF\xxx

# L16.2.8.4 Listing of Physical Examination

| Treatment | Patient<br>Randomization | | | |
|---|---|---|---|---|
| Group | Number | System | Visit 1 | Visit 3 /EOS |
| Test | XX-XXXX | General Appearance | Normal | Normal |
| | | Cardiovascular | | |
| | | Lungs and Thorax | | |
| | | Abdominal and Gastro-Enteric | | |
| | | etc | | |

Reference

Placebo

Test: Estradiol Vaginal Cream, USP, 0.01% (Teva Pharmaceuticals, USA)

Reference: Estrace® Cream (estradiol vaginal cream, USP, 0.01%; Warner Chilcott)

Placebo: Placebo cream (Teva Pharmaceuticals, USA)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\71436001\PDF\xxx

Created on: ddmmmyy hh:mm

# STATISTICAL ANALYSIS PLAN

# Estradiol Vaginal Cream, USP, 0.01%

Protocol / Study No. 71436001

#### 10. APPENDICIES

# Appendix A: Definitions and Severity Ratings For Signs and Symptoms

| Vaginal | Vaginal Dryness | |
|---|---|---|
| No lubric | No lubrication or secretions noted on perineum or after wiping; if sexually active loss of | |
| lubrication | lubrication during coitus. | |
| Score | Severity | Description |
| 0 | None | No noticeable lack of vaginal lubrication or secretions reported or |
| | | observed |
| 1 | Mild | Episodic loss of lubrication/secretions or noticed some reduction in |
| | | general secretions, does not interfere with daily activities |
| 2 | Moderate | Symptom present most of the time, and noticeable but overall is |
| | | tolerable and does not interfere with daily activities |
| 3 | Severe | Very minimal or no natural vaginal lubrication/secretions almost |
| | | all of the time and interferes with normal activities |

| Vaginal | Vaginal/Vulvar Irritation/Itching | |
|---|---|---|
| Scratchin | Scratching or sand paper type feeling in vaginal/vulvar area. May feel uncomfortable | |
| with clot | hing or unde | ergarments touching the perineum. |
| Score | Severity | Severity Description |
| 0 | None | No irritation or itching reported. |
| 1 | Mild | Occasional irritation/itching but does not interfere with daily |
| | | activities |
| 2 | Moderate | Frequent irritation/itching that can be uncomfortable but generally |
| | | does not interfere with daily activities |
| 3 | Severe | Very frequent or continuous irritation/itching of the vaginal area, |
| | | may interfere with daily activities. |

| Dysuria | | |
|---|---|---|
| Pain or discomfort during urination | | |
| Score | Severity | Description |
| 0 | None | No pain or discomfort during urination reported. |
| 1 | Mild | Occasional or slight discomfort during urination but tolerable |
| 2 | Moderate | Some discomfort during urination at least 50% of the time which |
| | | can be painful but overall tolerable. |
| 3 | Severe | Urination nearly always painful, usually intolerable and causing |
| | | disruption to daily activities |

# STATISTICAL ANALYSIS PLAN

# Estradiol Vaginal Cream, USP, 0.01%

# Protocol / Study No. 71436001

| Vaginal Pain during Sexual Activity | | |
|---|---|---|
| Suffers discomfort or pain during sexual activity that may be restrictive. | | |
| Score | Severity | Description |
| 0 | None | No discomfort or pain |
| 1 | Mild | Some feeling of vaginal soreness or pain, during or after sexual |
| | | activity. Does restrict frequency of or type of sexual activity. |
| 2 | Moderate | Vaginal pain during sexual activity such that frequency and type of sexual activity have been disrupted. Lubrication may be needed for penetration |
| 3 | Severe | Vaginal penetration very painful and impossible without vaginal lubrication. Discomfort such that frequency of sexual activity significantly reduced. |

| Vaginal bleeding during or after sexual activity | | |
|---|---|---|
| Score | Severity | Description |
| 0 | Absent | No vaginal bleeding observed |
| 1 | Present | Bleeding observed during or soon after vaginal activity |

At each visit each patient must also clearly identify which is the most bothersome sign/symptom to her, even if she rates two or more symptoms the same severity rating.